CLINICAL TRIAL: NCT01700439
Title: Multi-CenTer Experience With the Rapid Deployment EDWARDS INTUITY Valve System FOR Aortic Valve ReplaceMent
Brief Title: Surgical Treatment of Aortic Stenosis With a Next Generation, Rapid Deployment Surgical Aortic Valve
Acronym: TRANSFORM™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-02
Record Dates: First submitted 2012-09-19; First posted 2012-10-04 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Stenosis With Insufficiency; Regurgitation, Aortic Valve; Aortic Valve Incompetence
Keywords: Aortic valve; Heart valve; Tissue valve; Bioprosthesis; Valve disorder; Valve disease; Cardiac surgery; Less invasive cardiac surgery; Aortic valve stenosis; Aortic valve regurgitation; Bovine pericardium
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- EDWARDS INTUITY valve (Experimental): All subjects enrolled into the study are implanted with the EDWARDS INTUITY Valve System.
  Interventions: Device: EDWARDS INTUITY valve

INTERVENTIONS:
Device: EDWARDS INTUITY valve — Surgical replacement of the aortic valve with the EDWARDS INTUITY valve.

SUMMARY:
The purpose of the clinical study is to prove that the heart valve device is safe, effective, and performs as intended.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multi-center trial. Up to 950 subjects will be enrolled at up to 35 centers in the US. After replacement of their aortic heart valve with the EDWARDS INTUITY valve system, each patient will have routine follow-up tests at the following intervals: discharge, 3 months, 1 year, and annually thereafter for a minimum of five years.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria - Subjects will be required to meet all inclusion criteria:

  1. Male or female, age 18 years or older
  2. Has aortic stenosis or stenosis-insufficiency of an aortic valve requiring a planned replacement as indicated in the preoperative evaluation
  3. Is scheduled to undergo planned aortic valve replacement with or without concomitant coronary bypass surgery
  4. Provide written informed consent
  5. Geographically stable and agrees to attend follow-up assessments until all subjects have completed 5 years of follow up

Exclusion Criteria:

- Exclusion Criteria - Subjects will not be eligible for trial participation if any of the following criteria are present:

1. Pure aortic insufficiency
2. Requires emergency surgery
3. Previous aortic valve replacement
4. Had prior mitral, tricuspid or pulmonic valve surgery, which included implant of a bioprosthetic valve, mechanical valve, or annuloplasty ring that will remain in situ
5. Requires multiple valve replacement/repair
6. Requires a surgical procedure outside of the cardiac area (e.g., vascular endarterectomy, vascular bypass, tumor removal)
7. Aneurysm of the aortic root and/or ascending aorta requiring surgical intervention
8. Active endocarditis/myocarditis or endocarditis/ myocarditis within 3 months prior to the scheduled AVR surgery
9. Myocardial infarction (MI) within thirty (30) days prior to valve replacement surgery
10. Renal insufficiency as determined by creatinine ≥ 2.5 mg/dL at screening or end-stage renal disease requiring chronic dialysis
11. Hyperparathyroidism
12. MRI or CT-scan confirmed cerebrovascular accident (CVA), or transient ischemic attack (TIA) within 6 months (180 days) of the procedure
13. Presence of non-cardiac disease limiting life expectancy to less than 12 months
14. Hypertrophic obstructive cardiomyopathy (HOCM)
15. Left ventricular ejection fraction ≤ 25%
16. Documented history of substance (drug or alcohol) abuse within the last 5 years
17. Echocardiographic evidence of an intra-cardiac mass, thrombus, or vegetation
18. Hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 30 days prior to the procedure
19. Pregnancy, lactation, or planning to become pregnant;
20. Currently incarcerated or unable to give voluntary informed consent
21. Leucopenia (WBC < 3.5x 103/µL), or acute anemia (Hgb < 10.0 gm/dL or 6 mmol/L), or thrombocytopenia (platelet count < 50x 103/µL), or history of bleeding diathesis or coagulopathy
22. History of myxomatous disease/connective tissue disorders (e.g., Marfan's Syndrome)
23. Current or recent participation (within 6 weeks prior to surgery) in an investigational drug or device trial

    * Intra-operative Exclusion Criteria
24. Anatomic variances which contraindicate implant of the trial valve, such as:

    1. anomalous coronary arteries
    2. annular deformation or extensive calcification of the annulus or aortic root which cannot be removed
    3. significant calcium on the anterior mitral leaflet
    4. pronounced septal calcification
    5. position of coronary ostia relative to Model 8300ACD valve that would result in obstruction of blood flow
25. Available devices are not suitably sized for the subject's annulus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 934 (Actual)
Dates: Start 2012-09-26 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Barnhart, MD, Principal Investigator — Swedish Medical Center; Walter Randolph Chitwood, MD, Principal Investigator — East Carolina University
Locations (29):
- United States (29):
  - Keck Hospital of University of Southern California, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University, Palo Alto, California
  - Mercy General Hospital, Sacramento, California
  - Florida Hospital, Orlando, Florida
  - Northwestern University, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The University of Michigan Medical School, Ann Arbor, Michigan
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - North Shore Long Island Jewish Health System, Manhasset, New York
  - New York University Medical Center, New York, New York
  - Columbia University, New York, New York
  - Mission Hospital, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Pinnacle Health at Harrisburg Hospital, Harrisburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - St. Thomas Health, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Swedish Medical Center, Seattle, Washington
  - Aurora St Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

REFERENCES:
- [Result] Barnhart GR, Accola KD, Grossi EA, Woo YJ, Mumtaz MA, Sabik JF, Slachman FN, Patel HJ, Borger MA, Garrett HE Jr, Rodriguez E, McCarthy PM, Ryan WH, Duhay FG, Mack MJ, Chitwood WR Jr; TRANSFORM Trial Investigators. TRANSFORM (Multicenter Experience With Rapid Deployment Edwards INTUITY Valve System for Aortic Valve Replacement) US clinical trial: Performance of a rapid deployment aortic valve. J Thorac Cardiovasc Surg. 2017 Feb;153(2):241-251.e2. doi: 10.1016/j.jtcvs.2016.09.062. Epub 2016 Oct 15. PMID 27817951
- [Result] Romano MA, Koeckert M, Mumtaz MA, Slachman FN, Patel HJ, Chitwood WR Jr, Barnhart GR, Grossi EA; TRANSFORM Trial Investigators. Permanent Pacemaker Implantation After Rapid Deployment Aortic Valve Replacement. Ann Thorac Surg. 2018 Sep;106(3):685-690. doi: 10.1016/j.athoracsur.2018.03.055. Epub 2018 Apr 26. PMID 29705366

RESULTS

PARTICIPANT FLOW:
Groups:
- Edwards TRANSFORM Trial Cohort: Subjects who were enrolled in the TRANSFORM trial and were eligible to receive an INTUITY study surgical aortic heart valve.
Period: Overall Study
Arm/Group | Edwards TRANSFORM Trial Cohort
Started | 934
Study Valve Group | 885 (Received the Edwards INTUITY surgical aortic heart valve.)
Discharge | 925
3 Month | 862
1 Year | 842
2 Year | 795
3 Year | 720
4 Year | 667
5 Year | 577
6 Year | 357
7 Year | 164
8 Year | 40
Completed | 518
Not Completed | 416
Not completed — Lost to Follow-up | 47
Not completed — Withdrawal by Subject | 183
Not completed — Death | 186

BASELINE CHARACTERISTICS:
Groups:
- Edwards TRANSFORM Trial Cohort: Subjects who were enrolled in the TRANSFORM trial and were eligible to receive an Edwards INTUITY surgical aortic heart valve.
Arm/Group | Edwards TRANSFORM Trial Cohort
Number analyzed (Participants) | 934
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 336
  Male | 598
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 865
  Unknown or Not Reported | 65
Region of Enrollment [Number; unit: participants]
  United States | 934

OUTCOME MEASURES:

1. Primary Outcome: Number of Late Adverse Events Divided by Late Patient Years (Expressed as a Percentage) for the INTUTY Valve Implanted Cohort
Description: Late patient years are calculated from 31 days post-implant to the date of the last follow-up visits (or contact) or adverse events. Late Patient year calculation:[(Number of late adverse events/sum of late patient years) x 100]
Time Frame: Events occurring ≥ 31 days and up through 8 years post-implant
Population: The group of subjects that received the Edwards INTUITY surgical aortic heart valve.
Measure: Number; unit: Percentage of events/late patient years
Groups:
- Edwards INTUITY Surgical Aortic Heart Valve: Subjects who received an Edwards INTUITY surgical aortic heart valve.
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve
Number analyzed (Participants) | 885
Percentage of events/late patient years
  All cause mortality | 3.9
  Valve related mortality | 0.9
  Study valve reoperation | 0.6
  Study valve explant | 0.3
  Thromboembolism | 1.8
  Valve thrombosis | 0.0
  Endocarditis | 0.1
  All bleeding | 4.7
  Major bleeding | 2.4
  All paravalvular leak | 0.5
  Major paravalvular leak (PVL) | 0.3
  Hemolysis | 0.2
  Non-structural valve dysfunction other than PVL | 0.1
  Valve migration/embolization | 0.0
  Valve malposition | 0.0
  Valve instability | 0.0
  Valve dislodgement | 0.0
  Valve stenosis | 0.1
  Structural valve deterioration | 0.4
  Conduction defects | 0.4
  Conduction defects with permanent pacemaker | 0.1
  Conduction defects without permanent pacemaker | 0.3

2. Secondary Outcome: Percentage of Subjects With Edwards INTUITY Surgical Aortic Heart Valve Device Technical Success
Description: Device technical success is defined as the successful delivery and deployment of the aortic trial heart valve with maximum of two attempts and subject leaving the operating room (OR) with valve in place.
Time Frame: Day of procedure
Population: Patients who were eligible to receive an Edwards INTUITY surgical aortic heart valve.
Measure: Number; unit: Percentage of subjects
Arm/Group | Edwards TRANSFORM Trial Cohort
Number analyzed (Participants) | 934
Percentage of subjects | 94.8

3. Secondary Outcome: Percentage of Subjects With Edwards INTUITY Surgical Heart Valve Procedural Success
Description: Procedural success is defined as device technical success followed by the absence of adverse events resulting in device reoperation implant of permanent pacemaker (with baseline sinus rhythm and no other pre-existing conduction issues), or valve-related death within discharge or 10 days post index procedure, whichever comes first.
Time Frame: Day of procedure through discharge or 10 days post index procedure, whichever comes first.
Population: Patients who were eligible to receive an Edwards INTUITY surgical aortic heart valve.
Measure: Number; unit: Percentage of subjects
Arm/Group | Edwards TRANSFORM Trial Cohort
Number analyzed (Participants) | 934
Percentage of subjects | 94.4

4. Secondary Outcome: Average Amount of Time Subject Spent on Cardiopulmonary Bypass
Description: Surgical and hospitalization factors - Cardiopulmonary bypass time
Time Frame: Day of procedure
Population: The group of subjects that received the Edwards INTUITY surgical aortic heart valve.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Edwards INTUITY Surgical Aortic Heart Valve: Subjects who received an INTUITY study surgical aortic heart valve.
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve
Number analyzed (Participants) | 885
Minutes | 86.6 (37.4)

5. Secondary Outcome: Average Subject Time on Cardiopulmonary Cross Clamp
Description: Surgical and hospitalization factors - Cardiopulmonary cross clamp time
Time Frame: Day of procedure
Population: The group of subjects that received the Edwards INTUITY surgical aortic heart valve. Data is not available for one subject.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve
Number analyzed (Participants) | 884
Minutes | 65.4 (29.7)

6. Secondary Outcome: Average Number of Days Subjects Were in the Intensive Care Unit (ICU)
Description: Length of time surgical subjects were in the intensive care unit (ICU) after their heart valve replacement procedure.
Time Frame: Day of procedure through discharge from the hospital
Population: The group of subjects that received the Edwards INTUITY surgical aortic heart valve. Data is not available for 4 subjects.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve
Number analyzed (Participants) | 881
Days | 3.1 (3.7)

7. Secondary Outcome: Subject's New York Heart Association (NYHA) Classification Over Time
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life. Class I. Patients with cardiac disease but without resulting limitation of physical activity.
  Class II. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest.
  Class III. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Symptoms of heart failure or the anginal syndrome may be present even at rest.
Time Frame: Baseline, 3-months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8 Years
Population: This outcome is reported for subjects who received an Edwards INTUITY surgical aortic heart valve. Note that the number of participants analyzed is different from that in the participant flow as there was some missing data.
Measure: Count of Participants; unit: Participants
Groups:
- Edwards INTUITY Surgical Aortic Heart Valve - Class I; Edwards INTUITY Surgical Aortic Heart Valve - Class II; Edwards INTUITY Surgical Aortic Heart Valve - Class III; Edwards INTUITY Surgical Aortic Heart Valve - Class IV: Subjects who received an INTUITY study surgical aortic heart valve.
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve - Class I | Edwards INTUITY Surgical Aortic Heart Valve - Class II | Edwards INTUITY Surgical Aortic Heart Valve - Class III | Edwards INTUITY Surgical Aortic Heart Valve - Class IV
Number analyzed (Participants) | 885 | 885 | 885 | 885
Participants
  Baseline: number analyzed (Participants) | 882 | 882 | 882 | 882
  Baseline | 135 | 468 | 264 | 15
  3 months: number analyzed (Participants) | 839 | 839 | 839 | 839
  3 months | 671 | 148 | 20 | 0
  1 Year: number analyzed (Participants) | 814 | 814 | 814 | 814
  1 Year | 648 | 145 | 18 | 3
  2 Years: number analyzed (Participants) | 764 | 764 | 764 | 764
  2 Years | 606 | 133 | 22 | 3
  3 Years: number analyzed (Participants) | 693 | 693 | 693 | 693
  3 Years | 551 | 122 | 19 | 1
  4 Years: number analyzed (Participants) | 634 | 634 | 634 | 634
  4 Years | 487 | 123 | 21 | 3
  5 Years: number analyzed (Participants) | 543 | 543 | 543 | 543
  5 Years | 420 | 109 | 14 | 0
  6 Years: number analyzed (Participants) | 328 | 328 | 328 | 328
  6 Years | 251 | 63 | 14 | 0
  7 Years: number analyzed (Participants) | 144 | 144 | 144 | 144
  7 Years | 109 | 31 | 4 | 0
  8 Years: number analyzed (Participants) | 34 | 34 | 34 | 34
  8 Years | 28 | 5 | 1 | 0

8. Secondary Outcome: Subject's Average Mean Gradient Measurements Over Time
Description: Mean gradient is the average flow of blood through the aortic valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. In general, a higher value is considered worse, and a lower value is considered better but the value is dependent on the size and type of valve.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8-Years follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Edwards INTUITY Surgical Aortic Heart Valve - 19mm; Edwards INTUITY Surgical Aortic Heart Valve - 21mm; Edwards INTUITY Surgical Aortic Heart Valve - 23mm; Edwards INTUITY Surgical Aortic Heart Valve - 25mm; Edwards INTUITY Surgical Aortic Heart Valve - 27mm: Subjects who received an INTUITY study surgical aortic heart valve.
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve - 19mm | Edwards INTUITY Surgical Aortic Heart Valve - 21mm | Edwards INTUITY Surgical Aortic Heart Valve - 23mm | Edwards INTUITY Surgical Aortic Heart Valve - 25mm | Edwards INTUITY Surgical Aortic Heart Valve - 27mm
Number analyzed (Participants) | 49 | 179 | 291 | 261 | 105
mmHg
  Discharge: number analyzed (Participants) | 48 | 175 | 282 | 246 | 98
  Discharge | 17.7 (6.2) | 13.0 (4.1) | 12.3 (4.0) | 11.2 (3.7) | 9.7 (3.2)
  3 months: number analyzed (Participants) | 46 | 166 | 268 | 241 | 98
  3 months | 14.4 (4.4) | 11.1 (3.3) | 10.3 (3.5) | 9.7 (3.2) | 8.3 (2.5)
  1 Year: number analyzed (Participants) | 43 | 163 | 265 | 220 | 96
  1 Year | 13.9 (4.0) | 11.3 (3.6) | 10.0 (3.2) | 9.3 (3.0) | 8.1 (3.3)
  2 Years: number analyzed (Participants) | 43 | 144 | 249 | 211 | 89
  2 Years | 13.1 (4.5) | 11.1 (3.6) | 10.0 (3.7) | 9.3 (2.9) | 8.1 (3.6)
  3 Years: number analyzed (Participants) | 37 | 126 | 229 | 192 | 82
  3 Years | 13.7 (4.6) | 11.0 (4.3) | 10.0 (3.4) | 9.5 (3.5) | 7.9 (2.9)
  4 Years: number analyzed (Participants) | 34 | 113 | 201 | 175 | 80
  4 Years | 12.8 (3.8) | 10.8 (3.7) | 10.3 (6.7) | 9.5 (4.0) | 8.0 (3.7)
  5 Years: number analyzed (Participants) | 27 | 93 | 153 | 142 | 64
  5 Years | 12.4 (3.5) | 10.7 (3.9) | 10.0 (5.6) | 9.8 (6.5) | 7.9 (4.4)
  6 Years: number analyzed (Participants) | 22 | 55 | 94 | 80 | 32
  6 Years | 13.1 (3.9) | 10.5 (3.6) | 11.1 (6.4) | 9.3 (4.0) | 9.2 (6.5)
  7 Years: number analyzed (Participants) | 9 | 24 | 33 | 29 | 6
  7 Years | 12.1 (4.0) | 10.8 (3.1) | 12.8 (7.4) | 9.8 (4.0) | 7.7 (1.8)
  8 Years: number analyzed (Participants) | 1 | 7 | 10 | 6 | 2
  8 Years | 11.2 (0.0) | 13.2 (5.0) | 12.3 (8.3) | 12.9 (8.2) | 9.4 (2.2)

9. Secondary Outcome: Subject's Average Peak Gradient Measurements Over Time
Description: Peak gradient is the maximum value measured of flow of blood through the aortic valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. In general, a higher valve is considered worse, and a lower value is considered better, but the value is dependent on the size and type of valve.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8-Years follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve - 19mm | Edwards INTUITY Surgical Aortic Heart Valve - 21mm | Edwards INTUITY Surgical Aortic Heart Valve - 23mm | Edwards INTUITY Surgical Aortic Heart Valve - 25mm | Edwards INTUITY Surgical Aortic Heart Valve - 27mm
Number analyzed (Participants) | 49 | 179 | 291 | 261 | 105
mmHg
  Discharge: number analyzed (Participants) | 48 | 175 | 282 | 246 | 98
  Discharge | 32.8 (11.9) | 24.1 (7.9) | 22.9 (7.8) | 20.8 (6.8) | 17.9 (5.8)
  3 months: number analyzed (Participants) | 46 | 166 | 268 | 241 | 98
  3 months | 26.0 (8.0) | 19.9 (6.4) | 19.0 (6.5) | 17.6 (5.8) | 15.0 (4.4)
  1 Year: number analyzed (Participants) | 43 | 163 | 265 | 220 | 96
  1 Year | 25.0 (7.7) | 20.5 (6.5) | 18.2 (6.0) | 17.0 (5.7) | 14.6 (5.8)
  2 Years: number analyzed (Participants) | 43 | 144 | 249 | 211 | 89
  2 Years | 23.4 (7.9) | 20.2 (6.6) | 18.4 (6.8) | 17.0 (5.3) | 14.6 (6.2)
  3 Years: number analyzed (Participants) | 37 | 126 | 229 | 192 | 82
  3 Years | 24.7 (8.2) | 20.0 (7.8) | 18.5 (6.3) | 17.4 (6.3) | 14.5 (5.6)
  4 Years: number analyzed (Participants) | 34 | 113 | 201 | 175 | 80
  4 Years | 23.0 (6.6) | 19.8 (6.8) | 18.9 (10.4) | 17.6 (7.2) | 14.6 (6.6)
  5 Years: number analyzed (Participants) | 27 | 93 | 153 | 142 | 64
  5 Years | 22.7 (6.3) | 19.5 (7.0) | 18.4 (10.0) | 17.9 (10.7) | 14.5 (7.6)
  6 Years: number analyzed (Participants) | 22 | 55 | 94 | 80 | 32
  6 Years | 23.6 (6.1) | 19.1 (6.7) | 19.8 (9.4) | 17.1 (7.3) | 16.9 (10.9)
  7 Years: number analyzed (Participants) | 9 | 24 | 33 | 29 | 6
  7 Years | 22.1 (7.1) | 19.6 (5.9) | 23.5 (13.3) | 18.5 (7.7) | 14.6 (3.7)
  8 Years: number analyzed (Participants) | 1 | 7 | 10 | 6 | 2
  8 Years | 21.3 (0.0) | 24.4 (8.1) | 21.0 (12.6) | 22.7 (14.7) | 17.2 (3.6)

10. Secondary Outcome: Subject's Effective Orifice Area (EOA) Measurement Over Time
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the aortic valve. Effective orifice area is evaluated by echocardiography over time. In general, a higher value is considered better, and a lower value is considered worse, but the value is dependent on the size and type of valve.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8- Years follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Centimeters squared
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve - 19mm | Edwards INTUITY Surgical Aortic Heart Valve - 21mm | Edwards INTUITY Surgical Aortic Heart Valve - 23mm | Edwards INTUITY Surgical Aortic Heart Valve - 25mm | Edwards INTUITY Surgical Aortic Heart Valve - 27mm
Number analyzed (Participants) | 49 | 179 | 291 | 261 | 105
Centimeters squared
  Discharge: number analyzed (Participants) | 44 | 161 | 257 | 200 | 91
  Discharge | 1.1 (0.1) | 1.3 (0.2) | 1.7 (0.2) | 1.9 (0.2) | 2.2 (0.2)
  3 months: number analyzed (Participants) | 46 | 161 | 258 | 228 | 95
  3 months | 1.1 (0.1) | 1.3 (0.1) | 1.7 (0.2) | 1.9 (0.2) | 2.2 (0.2)
  1 Year: number analyzed (Participants) | 43 | 161 | 256 | 214 | 92
  1 Year | 1.1 (0.1) | 1.4 (0.1) | 1.7 (0.2) | 1.9 (0.2) | 2.2 (0.2)
  2 Years: number analyzed (Participants) | 42 | 142 | 240 | 201 | 85
  2 Years | 1.1 (0.1) | 1.4 (0.1) | 1.7 (0.2) | 1.9 (0.2) | 2.2 (0.2)
  3 Years: number analyzed (Participants) | 36 | 122 | 220 | 177 | 74
  3 Years | 1.1 (0.1) | 1.4 (0.1) | 1.7 (0.2) | 1.9 (0.2) | 2.1 (0.2)
  4 Years: number analyzed (Participants) | 33 | 111 | 193 | 167 | 76
  4 Years | 1.2 (0.1) | 1.4 (0.1) | 1.7 (0.2) | 1.9 (0.2) | 2.1 (0.3)
  5 Years: number analyzed (Participants) | 26 | 90 | 150 | 130 | 58
  5 Years | 1.2 (0.1) | 1.4 (0.2) | 1.7 (0.2) | 1.8 (0.2) | 2.1 (0.3)
  6 Years: number analyzed (Participants) | 22 | 53 | 88 | 78 | 31
  6 Years | 1.2 (0.1) | 1.4 (0.1) | 1.6 (0.2) | 1.9 (0.2) | 2.0 (0.3)
  7 Years: number analyzed (Participants) | 9 | 23 | 32 | 27 | 4
  7 Years | 1.2 (0.1) | 1.4 (0.1) | 1.6 (0.3) | 1.8 (0.3) | 2.1 (0.1)
  8 Years: number analyzed (Participants) | 1 | 6 | 9 | 5 | 2
  8 Years | 1.1 (0.0) | 1.4 (0.1) | 1.6 (0.3) | 1.7 (0.3) | 2.1 (0.1)

11. Secondary Outcome: Subject's Effective Orifice Area Index (EOAI) Measurement Over Time
Description: Effective orifice area index represents the minimal cross-sectional area of the blood flow downstream of the mitral valve divided by the person's body surface area. Effective orifice area index is evaluated by echocardiography over time. In general, a higher value is considered better, and a lower value is considered worse, but the value is dependent on the size of the patient and the size and type of valve.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8- Years follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: centimeters squared/meters squared
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve - 19mm | Edwards INTUITY Surgical Aortic Heart Valve - 21mm | Edwards INTUITY Surgical Aortic Heart Valve - 23mm | Edwards INTUITY Surgical Aortic Heart Valve - 25mm | Edwards INTUITY Surgical Aortic Heart Valve - 27mm
Number analyzed (Participants) | 49 | 179 | 291 | 261 | 105
centimeters squared/meters squared
  Discharge: number analyzed (Participants) | 44 | 160 | 256 | 199 | 91
  Discharge | 0.6 (0.1) | 0.7 (0.1) | 0.8 (0.1) | 0.9 (0.1) | 1.0 (0.1)
  3 months: number analyzed (Participants) | 46 | 161 | 257 | 228 | 95
  3 months | 0.7 (0.1) | 0.7 (0.1) | 0.8 (0.1) | 0.9 (0.1) | 1.0 (0.1)
  1 Year: number analyzed (Participants) | 43 | 161 | 256 | 211 | 92
  1 Year | 0.7 (0.1) | 0.7 (0.1) | 0.8 (0.1) | 0.9 (0.1) | 1.0 (0.1)
  2 Years: number analyzed (Participants) | 42 | 142 | 239 | 198 | 85
  2 Years | 0.7 (0.1) | 0.7 (0.1) | 0.8 (0.1) | 0.9 (0.1) | 1.0 (0.1)
  3 Years: number analyzed (Participants) | 35 | 122 | 220 | 177 | 74
  3 Years | 0.7 (0.1) | 0.7 (0.1) | 0.8 (0.1) | 0.9 (0.1) | 1.0 (0.1)
  4 Years: number analyzed (Participants) | 33 | 111 | 193 | 167 | 76
  4 Years | 0.7 (0.1) | 0.8 (0.1) | 0.8 (0.1) | 0.9 (0.1) | 1.0 (0.1)
  5 Years: number analyzed (Participants) | 26 | 90 | 150 | 129 | 58
  5 Years | 0.7 (0.1) | 0.7 (0.1) | 0.8 (0.1) | 0.9 (0.1) | 1.0 (0.1)
  6 Years: number analyzed (Participants) | 22 | 51 | 87 | 77 | 31
  6 Years | 0.7 (0.1) | 0.7 (0.1) | 0.8 (0.1) | 0.9 (0.1) | 0.9 (0.2)
  7 Years: number analyzed (Participants) | 9 | 23 | 32 | 27 | 4
  7 Years | 0.7 (0.1) | 0.7 (0.1) | 0.8 (0.2) | 0.9 (0.2) | 1.0 (0.1)
  8 Years: number analyzed (Participants) | 1 | 6 | 9 | 5 | 2
  8 Years | 0.6 (0.0) | 0.7 (0.1) | 0.8 (0.2) | 0.8 (0.2) | 1.0 (0.1)

12. Secondary Outcome: Subject's Performance Index Measurement Over Time
Description: Performance index is defined as the subject's effective orifice area (the cross-sectional area of the blood flow downstream of the aortic valve) divided by the subject's native orifice area. Performance Index is evaluated by echocardiography over time and are dependent on the size and type of the valve. In general, a higher value is considered better, and a lower value is considered worse, but the value is dependent on the size of the patient and the size and type of valve.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8- Years follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Centimeters squared/meters squared
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve - 19mm | Edwards INTUITY Surgical Aortic Heart Valve - 21mm | Edwards INTUITY Surgical Aortic Heart Valve - 23mm | Edwards INTUITY Surgical Aortic Heart Valve - 25mm | Edwards INTUITY Surgical Aortic Heart Valve - 27mm
Number analyzed (Participants) | 49 | 179 | 291 | 261 | 105
Centimeters squared/meters squared
  Discharge: number analyzed (Participants) | 44 | 161 | 257 | 200 | 91
  Discharge | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.8 (0.1)
  3 months: number analyzed (Participants) | 46 | 161 | 258 | 228 | 95
  3 months | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.8 (0.1)
  1 Year: number analyzed (Participants) | 43 | 161 | 256 | 214 | 92
  1 Year | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.8 (0.1)
  2 Years: number analyzed (Participants) | 42 | 142 | 240 | 201 | 85
  2 Years | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.8 (0.1)
  3 Years: number analyzed (Participants) | 36 | 122 | 220 | 177 | 74
  3 Years | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.8 (0.1)
  4 Years: number analyzed (Participants) | 33 | 111 | 193 | 167 | 76
  4 Years | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.8 (0.1)
  5 Years: number analyzed (Participants) | 26 | 90 | 150 | 130 | 58
  5 Years | 1.0 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.9 (0.1) | 0.8 (0.1)
  6 Years: number analyzed (Participants) | 22 | 53 | 88 | 78 | 31
  6 Years | 1.0 (0.1) | 0.9 (0.1) | 0.8 (0.1) | 0.9 (0.1) | 0.8 (0.1)
  7 Years: number analyzed (Participants) | 9 | 23 | 32 | 27 | 4
  7 Years | 1.0 (0.1) | 0.9 (0.1) | 0.8 (0.1) | 0.9 (0.1) | 0.8 (0.0)
  8 Years: number analyzed (Participants) | 1 | 6 | 9 | 5 | 2
  8 Years | 0.9 (0.0) | 0.9 (0.1) | 0.8 (0.2) | 0.8 (0.1) | 0.8 (0.0)

13. Secondary Outcome: Subject's Cardiac Output Measurement at Over Time
Description: Cardiac output is the amount of blood the heart pumps through the circulatory system in a minute. Cardiac output is evaluated by echocardiography over time. Normal cardiac output in healthy volunteers over 60 years of age was reported between 3.1 and 6.4 liters per minute. In general, a higher value is considered better, and a lower value is considered worse.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8- Years follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters/minutes
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve - 19mm | Edwards INTUITY Surgical Aortic Heart Valve - 21mm | Edwards INTUITY Surgical Aortic Heart Valve - 23mm | Edwards INTUITY Surgical Aortic Heart Valve - 25mm | Edwards INTUITY Surgical Aortic Heart Valve - 27mm
Number analyzed (Participants) | 49 | 179 | 291 | 261 | 105
Liters/minutes
  Discharge: number analyzed (Participants) | 44 | 162 | 261 | 207 | 93
  Discharge | 4.3 (0.9) | 4.6 (0.9) | 5.4 (1.1) | 5.6 (1.1) | 5.9 (1.3)
  3 months: number analyzed (Participants) | 46 | 161 | 260 | 231 | 100
  3 months | 4.3 (0.7) | 4.4 (0.8) | 5.0 (0.9) | 5.2 (1.0) | 5.4 (1.1)
  1 Year: number analyzed (Participants) | 45 | 161 | 259 | 220 | 93
  1 Year | 4.3 (0.9) | 4.4 (1.0) | 4.9 (0.9) | 5.1 (1.0) | 5.5 (1.2)
  2 Years: number analyzed (Participants) | 42 | 144 | 245 | 207 | 87
  2 Years | 4.1 (0.8) | 4.3 (0.8) | 4.9 (0.9) | 5.0 (1.0) | 5.3 (1.0)
  3 Years: number analyzed (Participants) | 36 | 124 | 226 | 185 | 76
  3 Years | 4.0 (0.7) | 4.3 (0.9) | 4.9 (0.9) | 5.1 (1.0) | 5.2 (1.1)
  4 Years: number analyzed (Participants) | 33 | 111 | 198 | 172 | 78
  4 Years | 4.1 (0.8) | 4.1 (0.8) | 4.9 (1.0) | 5.1 (1.0) | 5.2 (1.1)
  5 Years: number analyzed (Participants) | 26 | 92 | 157 | 141 | 61
  5 Years | 4.2 (0.7) | 4.3 (0.9) | 4.8 (1.0) | 5.0 (1.1) | 5.2 (0.9)
  6 Years: number analyzed (Participants) | 22 | 53 | 91 | 87 | 32
  6 Years | 4.3 (0.7) | 4.2 (0.9) | 4.9 (1.1) | 5.0 (1.1) | 5.3 (1.2)
  7 Years: number analyzed (Participants) | 9 | 23 | 34 | 27 | 4
  7 Years | 3.9 (0.6) | 4.2 (0.8) | 5.0 (1.0) | 5.1 (1.1) | 5.0 (0.9)
  8 Years: number analyzed (Participants) | 1 | 6 | 9 | 5 | 2
  8 Years | 2.9 (0.0) | 4.9 (1.6) | 5.4 (1.3) | 4.9 (1.3) | 5.5 (1.3)

14. Secondary Outcome: Subject's Cardiac Index Measurement Over Time
Description: Hemodynamic performance - Cardiac index (CI) evaluated by echocardiography. Cardiac index is an assessment of the cardiac output value based on the patient's size. To obtain the cardiac index, divide the cardiac output by the person's body surface area (BSA). Cardiac Index is a useful marker of how well the heart is functioning as a pump by directly correlating the volume of blood pumped by the heart with an individual's body surface area. Normal cardiac output index in healthy volunteers over 60 years of age was reported between 1.1 and 3.2 L/min/m^2. In general, a higher value is considered better, and a lower value is considered worse, but the value is dependent on the size of the patient.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8- Years follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters/minutes/meters squared
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve - 19mm | Edwards INTUITY Surgical Aortic Heart Valve - 21mm | Edwards INTUITY Surgical Aortic Heart Valve - 23mm | Edwards INTUITY Surgical Aortic Heart Valve - 25mm | Edwards INTUITY Surgical Aortic Heart Valve - 27mm
Number analyzed (Participants) | 49 | 179 | 291 | 261 | 105
Liters/minutes/meters squared
  Discharge: number analyzed (Participants) | 44 | 161 | 260 | 206 | 93
  Discharge | 2.5 (0.5) | 2.4 (0.5) | 2.7 (0.5) | 2.6 (0.6) | 2.7 (0.6)
  3 months: number analyzed (Participants) | 46 | 161 | 259 | 231 | 100
  3 months | 2.6 (0.5) | 2.4 (0.4) | 2.5 (0.5) | 2.5 (0.5) | 2.5 (0.5)
  1 Year: number analyzed (Participants) | 45 | 161 | 259 | 216 | 93
  1 Year | 2.5 (0.6) | 2.4 (0.5) | 2.4 (0.4) | 2.4 (0.5) | 2.5 (0.6)
  2 Years: number analyzed (Participants) | 42 | 144 | 244 | 204 | 87
  2 Years | 2.4 (0.5) | 2.3 (0.4) | 2.4 (0.5) | 2.4 (0.5) | 2.4 (0.4)
  3 Years: number analyzed (Participants) | 35 | 124 | 226 | 185 | 76
  3 Years | 2.3 (0.4) | 2.3 (0.5) | 2.4 (0.4) | 2.4 (0.5) | 2.4 (0.5)
  4 Years: number analyzed (Participants) | 33 | 111 | 198 | 172 | 78
  4 Years | 2.3 (0.5) | 2.3 (0.4) | 2.4 (0.5) | 2.4 (0.5) | 2.4 (0.5)
  5 Years: number analyzed (Participants) | 26 | 92 | 157 | 140 | 61
  5 Years | 2.4 (0.5) | 2.3 (0.5) | 2.4 (0.5) | 2.3 (0.5) | 2.4 (0.4)
  6 Years: number analyzed (Participants) | 22 | 51 | 90 | 86 | 32
  6 Years | 2.5 (0.5) | 2.3 (0.4) | 2.4 (0.6) | 2.4 (0.6) | 2.4 (0.6)
  7 Years: number analyzed (Participants) | 9 | 23 | 34 | 27 | 4
  7 Years | 2.3 (0.4) | 2.2 (0.4) | 2.5 (0.5) | 2.4 (0.5) | 2.3 (0.3)
  8 Years: number analyzed (Participants) | 1 | 6 | 9 | 5 | 2
  8 Years | 1.5 (0.0) | 2.6 (0.9) | 2.6 (0.6) | 2.4 (0.6) | 2.8 (0.2)

15. Secondary Outcome: Amount of Aortic Valvular Regurgitation in Subjects Over Time by Valve Size
Description: Valvular regurgitation occurs when the valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation and 4 represents severe regurgitation. Higher numbers on the scale show a worsening outcome.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8- Years follow-up
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve - 19mm | Edwards INTUITY Surgical Aortic Heart Valve - 21mm | Edwards INTUITY Surgical Aortic Heart Valve - 23mm | Edwards INTUITY Surgical Aortic Heart Valve - 25mm | Edwards INTUITY Surgical Aortic Heart Valve - 27mm
Number analyzed (Participants) | 49 | 179 | 291 | 261 | 105
Participants
  Discharge: number analyzed (Participants) | 48 | 176 | 283 | 250 | 102
  Discharge: None (0)/Trival (+1) | 46 | 171 | 266 | 235 | 97
  Discharge: Mild (+2) | 2 | 3 | 12 | 13 | 3
  Discharge: Moderate (+3) | 0 | 2 | 4 | 0 | 2
  Discharge: Severe (+4) | 0 | 0 | 1 | 2 | 0
  3 months: number analyzed (Participants) | 45 | 168 | 266 | 244 | 105
  3 months: None (0)/Trival (+1) | 43 | 156 | 245 | 219 | 97
  3 months: Mild (+2) | 2 | 12 | 16 | 18 | 4
  3 months: Moderate (+3) | 0 | 0 | 4 | 6 | 4
  3 months: Severe (+4) | 0 | 0 | 1 | 1 | 0
  1 Year: number analyzed (Participants) | 45 | 166 | 268 | 224 | 96
  1 Year: None (0)/Trival (+1) | 40 | 156 | 245 | 200 | 89
  1 Year: Mild (+2) | 5 | 9 | 18 | 21 | 5
  1 Year: Moderate (+3) | 0 | 1 | 5 | 2 | 1
  1 Year: Severe (+4) | 0 | 0 | 0 | 1 | 1
  2 Years: number analyzed (Participants) | 43 | 146 | 252 | 217 | 92
  2 Years: None (0)/Trival (+1) | 38 | 138 | 229 | 193 | 86
  2 Years: Mild (+2) | 5 | 8 | 19 | 23 | 4
  2 Years: Moderate (+3) | 0 | 0 | 4 | 0 | 2
  2 Years: Severe (+4) | 0 | 0 | 0 | 1 | 0
  3 Years: number analyzed (Participants) | 38 | 127 | 232 | 197 | 86
  3 Years: None (0)/Trival (+1) | 33 | 120 | 211 | 179 | 79
  3 Years: Mild (+2) | 5 | 7 | 18 | 18 | 5
  3 Years: Moderate (+3) | 0 | 0 | 3 | 0 | 2
  3 Years: Severe (+4) | 0 | 0 | 0 | 0 | 0
  4 Years: number analyzed (Participants) | 35 | 113 | 209 | 179 | 82
  4 Years: None (0)/Trival (+1) | 31 | 104 | 191 | 160 | 77
  4 Years: Mild (+2) | 4 | 9 | 17 | 19 | 5
  4 Years: Moderate (+3) | 0 | 0 | 1 | 0 | 0
  4 Years: Severe (+4) | 0 | 0 | 0 | 0 | 0
  5 Years: number analyzed (Participants) | 28 | 94 | 161 | 149 | 66
  5 Years: None (0)/Trival (+1) | 26 | 87 | 146 | 129 | 61
  5 Years: Mild (+2) | 2 | 7 | 15 | 18 | 4
  5 Years: Moderate (+3) | 0 | 0 | 0 | 1 | 1
  5 Years: Severe (+4) | 0 | 0 | 0 | 1 | 0
  6 Years: number analyzed (Participants) | 22 | 55 | 97 | 88 | 33
  6 Years: None (0)/Trival (+1) | 20 | 53 | 87 | 78 | 31
  6 Years: Mild (+2) | 2 | 2 | 9 | 10 | 2
  6 Years: Moderate (+3) | 0 | 0 | 1 | 0 | 0
  6 Years: Severe (+4) | 0 | 0 | 0 | 0 | 0
  7 Years: number analyzed (Participants) | 9 | 26 | 35 | 29 | 6
  7 Years: None (0)/Trival (+1) | 7 | 25 | 30 | 22 | 6
  7 Years: Mild (+2) | 2 | 1 | 5 | 6 | 0
  7 Years: Moderate (+3) | 0 | 0 | 0 | 1 | 0
  7 Years: Severe (+4) | 0 | 0 | 0 | 0 | 0
  8 Years: number analyzed (Participants) | 1 | 7 | 10 | 6 | 2
  8 Years: None (0)/Trival (+1) | 1 | 6 | 10 | 4 | 2
  8 Years: Mild (+2) | 0 | 1 | 0 | 2 | 0
  8 Years: Moderate (+3) | 0 | 0 | 0 | 0 | 0
  8 Years: Severe (+4) | 0 | 0 | 0 | 0 | 0

16. Other Pre Specified Outcome: Subject's Average Score at Baseline and 1 Year on the Quality of Life Survey
Description: The Medical Outcomes Study Short-Form 12 (SF-12) - physical and metal states. The SF-12 questionnaire scale ranges from 100, which reflects the best health status to 0, which reflects the worst health status.
Time Frame: Baseline and one year follow-up
Population: This outcome is reported for subjects who received an Edwards INTUITY surgical aortic heart valve where data is available at both the baseline and 1 year follow-up visits. Note that the number of participants analyzed is different from that in the participant flow as there was some missing data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve
Number analyzed (Participants) | 524
Units on a scale
  Mental Health - Baseline | 51.3 (9.9)
  Mental Health - 1 year follow-up | 54.3 (8.5)
  Physical Health - Baseline | 41.8 (10.2)
  Physical Health - 1 year follow-up | 47.6 (9.7)

17. Other Pre Specified Outcome: Subject's Average White Blood Cell Count Over Time
Description: Laboratory analysis of White Blood Cell (WBC) count on blood drawn from subject; WBC fight infection. The normal reference range for WBC count is 4.5 to 10 10^3 cells/microliters. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8- Years follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliters
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve
Number analyzed (Participants) | 885
10^3 cells/microliters
  Discharge: number analyzed (Participants) | 878
  Discharge | 9.54 (3.0)
  3 months: number analyzed (Participants) | 825
  3 months | 7.27 (2.5)
  1 Year: number analyzed (Participants) | 800
  1 Year | 7.31 (2.8)
  2 Years: number analyzed (Participants) | 751
  2 Years | 7.47 (4.5)
  3 Years: number analyzed (Participants) | 690
  3 Years | 7.47 (5.7)
  4 Years: number analyzed (Participants) | 629
  4 Years | 7.41 (3.0)
  5 Years: number analyzed (Participants) | 512
  5 Years | 7.37 (3.6)
  6 Years: number analyzed (Participants) | 290
  6 Years | 7.47 (6.1)
  7 Years: number analyzed (Participants) | 114
  7 Years | 8.05 (9.8)
  8 Years: number analyzed (Participants) | 29
  8 Years | 14.0 (36.8)

18. Other Pre Specified Outcome: Subject's Average Red Blood Cell Count Over Time
Description: The red blood cell (RBC) count is a test that measures the number of oxygen-carrying blood cells in your blood. The red blood cell count normal range for women is 4.2 to 5.4 10^6 cells/microliters and for men is 4.7 to 6.1 10^6 cells/microliters. A high red blood cell count may indicate that you have a condition that's preventing you from getting enough oxygen. A low RBC may be caused by an infection, or a medical condition related to anemia. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8- Years follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliters
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve
Number analyzed (Participants) | 885
10^6 cells/microliters
  Discharge: number analyzed (Participants) | 878
  Discharge | 3.31 (0.5)
  3 months: number analyzed (Participants) | 825
  3 months | 4.51 (0.5)
  1 Year: number analyzed (Participants) | 800
  1 Year | 4.46 (0.5)
  2 Years: number analyzed (Participants) | 751
  2 Years | 4.45 (0.5)
  3 Years: number analyzed (Participants) | 690
  3 Years | 4.46 (0.5)
  4 Years: number analyzed (Participants) | 627
  4 Years | 4.44 (0.5)
  5 Years: number analyzed (Participants) | 510
  5 Years | 4.43 (0.6)
  6 Years: number analyzed (Participants) | 289
  6 Years | 4.38 (0.5)
  7 Years: number analyzed (Participants) | 113
  7 Years | 4.33 (0.6)
  8 Years: number analyzed (Participants) | 29
  8 Years | 4.28 (0.7)

19. Other Pre Specified Outcome: Subject's Average Hematocrit Percentage Over Time
Description: Laboratory Analysis of Hematocrit Percentage on blood drawn from subjects. A hematocrit test measures the proportion of red blood cells in your blood. Red blood cells carry oxygen throughout your body. Having too few or too many red blood cells can be a sign of certain diseases. Normal hematocrit ranges for adult females are 36% to 44% and for adult males are 41% to 50%. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8- Years follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of RBC
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve
Number analyzed (Participants) | 885
Percentage of RBC
  Discharge: number analyzed (Participants) | 878
  Discharge | 29.94 (4.0)
  3 months: number analyzed (Participants) | 825
  3 months | 39.28 (4.2)
  1 Year: number analyzed (Participants) | 800
  1 Year | 40.25 (4.4)
  2 Years: number analyzed (Participants) | 751
  2 Years | 40.30 (4.4)
  3 Years: number analyzed (Participants) | 689
  3 Years | 40.42 (4.1)
  4 Years: number analyzed (Participants) | 629
  4 Years | 40.40 (4.2)
  5 Years: number analyzed (Participants) | 512
  5 Years | 40.66 (4.5)
  6 Years: number analyzed (Participants) | 291
  6 Years | 40.41 (4.4)
  7 Years: number analyzed (Participants) | 113
  7 Years | 40.00 (4.8)
  8 Years: number analyzed (Participants) | 29
  8 Years | 39.31 (5.4)

20. Other Pre Specified Outcome: Subject's Average Hemoglobin Percentage Over Time
Description: Laboratory Analysis of Hemoglobin Count on blood drawn from subjects. Hemoglobin is an oxygen-carrying protein in red blood cells. In males, a healthy hemoglobin level is between 13.2 and 16.6 g/dL. In females, a hemoglobin count of between 11.6 and 15 g/dL is considered normal and healthy. In general, results either lower or higher than the normal range can indicate something is wrong.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8- Years follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve
Number analyzed (Participants) | 885
g/dL
  Discharge: number analyzed (Participants) | 878
  Discharge | 9.95 (1.4)
  3 months: number analyzed (Participants) | 826
  3 months | 12.82 (1.6)
  1 Year: number analyzed (Participants) | 800
  1 Year | 13.33 (1.6)
  2 Years: number analyzed (Participants) | 752
  2 Years | 13.37 (1.6)
  3 Years: number analyzed (Participants) | 690
  3 Years | 13.42 (1.6)
  4 Years: number analyzed (Participants) | 630
  4 Years | 13.39 (1.6)
  5 Years: number analyzed (Participants) | 511
  5 Years | 13.22 (2.2)
  6 Years: number analyzed (Participants) | 291
  6 Years | 13.20 (1.8)
  7 Years: number analyzed (Participants) | 115
  7 Years | 13.10 (1.8)
  8 Years: number analyzed (Participants) | 30
  8 Years | 12.87 (1.9)

21. Other Pre Specified Outcome: Subject's Average Plasma Free Hemoglobin Over Time
Description: Laboratory Analysis of Plasma Free Hemoglobin (Hgb) of blood drawn from subject. This blood test measures the level of free hemoglobin in the plasma (liquid portion of the blood). The reference range for plasma free hemoglobin is 0.0 to 15.2 mg/dL. In general, values higher than this can indicate something is wrong.
Time Frame: Discharge, 3 months, 1-, 2-, 3-, 4-, 5-, 6-, 7-, and 8- Years follow-up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve
Number analyzed (Participants) | 885
mg/dL
  Discharge: number analyzed (Participants) | 737
  Discharge | 11.89 (14.6)
  3 months: number analyzed (Participants) | 708
  3 months | 13.12 (13.5)
  1 Year: number analyzed (Participants) | 640
  1 Year | 12.08 (12.9)
  2 Years: number analyzed (Participants) | 518
  2 Years | 12.06 (13.5)
  3 Years: number analyzed (Participants) | 457
  3 Years | 11.90 (15.7)
  4 Years: number analyzed (Participants) | 411
  4 Years | 11.88 (14.5)
  5 Years: number analyzed (Participants) | 314
  5 Years | 12.73 (16.9)
  6 Years: number analyzed (Participants) | 155
  6 Years | 16.32 (14.4)
  7 Years: number analyzed (Participants) | 55
  7 Years | 18.43 (14.9)
  8 Years: number analyzed (Participants) | 11
  8 Years | 22.61 (11.4)

ADVERSE EVENTS:
Time Frame: Events occurring from the day of aortic heart valve surgery up through 8 years post implant.
Groups:
- Edwards TRANSFORM INTUITY Aortic Valve Study Cohort: The data from the 885 subjects who received the investigational Edwards INTUITY surgical aortic heart valve.
- Commercially Available Aortic Valve Study Cohort: The data from the 49 subjects who received an alternate FDA approved surgical aortic heart valve.
Arm/Group | Edwards TRANSFORM INTUITY Aortic Valve Study Cohort | Commercially Available Aortic Valve Study Cohort
All-Cause Mortality (participants affected / at risk) | 178/885 | 8/49
Serious Adverse Events (participants affected / at risk) | 756/885 | 37/49
Other Adverse Events (participants affected / at risk) | 868/885 | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edwards TRANSFORM INTUITY Aortic Valve Study Cohort (N=885) | Commercially Available Aortic Valve Study Cohort (N=49)
ANEMIA - BLEEDING RELATED - MAJOR (Blood and lymphatic system disorders) | 31 | 4
ANEMIA - BLEEDING RELATED - MINOR (Blood and lymphatic system disorders) | 45 | 5
ANEMIA - NON-BLEEDING RELATED (Blood and lymphatic system disorders) | 28 | 1
BLEEDING - CARDIOVASCULAR - MAJOR (Blood and lymphatic system disorders) | 20 | 3
BLEEDING - CARDIOVASCULAR - MINOR (Blood and lymphatic system disorders) | 12 | 1
BLEEDING - GASTROINTESTINAL LOWER - MAJOR (Blood and lymphatic system disorders) | 16 | 1
BLEEDING - GASTROINTESTINAL LOWER - MINOR (Blood and lymphatic system disorders) | 17 | 0
BLEEDING - GASTROINTESTINAL UPPER - MAJOR (Blood and lymphatic system disorders) | 18 | 0
BLEEDING - GASTROINTESTINAL UPPER - MINOR (Blood and lymphatic system disorders) | 10 | 2
BLEEDING - GENITOURINARY - MAJOR (Blood and lymphatic system disorders) | 4 | 1
BLEEDING - GENITOURINARY - MINOR (Blood and lymphatic system disorders) | 7 | 0
BLEEDING - MUSCULOSKELETAL/DERMATOLOGICAL - MAJOR (E.G. ECCHYMOSIS) (Blood and lymphatic system disorders) | 1 | 0
BLEEDING - MUSCULOSKELETAL/DERMATOLOGICAL - MINOR (E.G. ECCHYMOSIS) (Blood and lymphatic system disorders) | 5 | 2
BLEEDING - NEUROLOGICAL - MAJOR (E.G. CVA) (Blood and lymphatic system disorders) | 15 | 0
BLEEDING - NEUROLOGICAL - MINOR (E.G. CVA) (Blood and lymphatic system disorders) | 5 | 0
BLEEDING - PERIPHERAL VASCULAR - MAJOR (E.G. NOSEBLEEDS; HEMATOMAS) (Blood and lymphatic system disorders) | 4 | 0
BLEEDING - PULMONARY/RESPIRATORY - MAJOR (E.G. HEMOTHORAX) (Blood and lymphatic system disorders) | 3 | 0
BLEEDING - PULMONARY/RESPIRATORY - MINOR (E.G. HEMOTHORAX) (Blood and lymphatic system disorders) | 2 | 0
BLOOD SEPSIS (Blood and lymphatic system disorders) | 49 | 1
BLOOD/LYMPHATIC - OTHER (Blood and lymphatic system disorders) | 23 | 2
THROMBOCYTOPENIA - HEPARIN INDUCED (HIT) (Blood and lymphatic system disorders) | 5 | 0
THROMBOCYTOPENIA - NON-HEPARIN INDUCED (Blood and lymphatic system disorders) | 23 | 2
ANGINA, STABLE (Cardiac disorders) | 21 | 0
ANGINA, UNSTABLE (Cardiac disorders) | 22 | 0
AORTIC DISSECTION (Cardiac disorders) | 3 | 1
ARRHYTHMIA - ATRIAL FLUTTER (Cardiac disorders) | 37 | 0
ARRHYTHMIA - AV BLOCK - 1ST DEGREE (Cardiac disorders) | 4 | 0
ARRHYTHMIA - AV BLOCK - 2ND DEGREE (Cardiac disorders) | 17 | 1
ARRHYTHMIA - AV BLOCK - 3RD DEGREE (Cardiac disorders) | 94 | 2
ARRHYTHMIA - BRADYCARDIA (Cardiac disorders) | 28 | 1
ARRHYTHMIA - BUNDLE BRANCH BLOCK - LEFT (Cardiac disorders) | 9 | 0
ARRHYTHMIA - BUNDLE BRANCH BLOCK - RIGHT (Cardiac disorders) | 2 | 0
ARRHYTHMIA - OTHER (Cardiac disorders) | 34 | 2
ARRHYTHMIA - PACEMAKER/ICD MALFUNCTION (Cardiac disorders) | 2 | 0
ARRHYTHMIA - PAROXYSMAL ATRIAL FIBRILLATION (PAF) (Cardiac disorders) | 91 | 12
ARRHYTHMIA - PAROXYSMAL ATRIAL TACHYCARDIA (PAT) (Cardiac disorders) | 1 | 0
ARRHYTHMIA - PERMANENT ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 0
ARRHYTHMIA - PERSISTENT ATRIAL FIBRILLATION (Cardiac disorders) | 68 | 5
ARRHYTHMIA - SUPRAVENTRICULAR TACHYCARDIA (SVT) (Cardiac disorders) | 5 | 0
ARRHYTHMIA - TACHY-BRADYCARDIA (Cardiac disorders) | 12 | 1
ARRHYTHMIA - TACHYCARDIA - NON-VENTRICULAR (Cardiac disorders) | 5 | 0
ARRHYTHMIA - TACHYCARDIA - VENTRICULAR (Cardiac disorders) | 8 | 1
ARRHYTHMIA - VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 | 1
CARDIAC ARREST (Cardiac disorders) | 27 | 2
CARDIAC DECOMPENSATION (Cardiac disorders) | 2 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 14 | 4
CARDIOVASCULAR - OTHER (Cardiac disorders) | 105 | 4
CORONARY ARTERY OSTIAL OBSTRUCTION (Cardiac disorders) | 3 | 1
ENDOCARDITIS (Cardiac disorders) | 11 | 1
HEART FAILURE - ACUTE (Cardiac disorders) | 64 | 4
HEART FAILURE - CHRONIC (CHF) (Cardiac disorders) | 42 | 1
HYPERTENSION - SYSTEMIC (Cardiac disorders) | 16 | 0
HYPOTENSION (Cardiac disorders) | 25 | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 34 | 1
PERFORATION - VENTRICULAR (Cardiac disorders) | 1 | 0
PERICARDIAL EFFUSION - MAJOR (Cardiac disorders) | 14 | 3
PERICARDIAL EFFUSION - MINOR (Cardiac disorders) | 4 | 0
PERICARDIAL TAMPONADE (Cardiac disorders) | 4 | 2
PERICARDITIS (Cardiac disorders) | 5 | 0
REGURGITATION - AORTIC-CENTRAL/TRANSVALVULAR +4 (Cardiac disorders) | 2 | 0
REGURGITATION - MITRAL-CENTRAL/TRANSVALVULAR +3 (Cardiac disorders) | 2 | 0
REGURGITATION - MITRAL-CENTRAL/TRANSVALVULAR +4 (Cardiac disorders) | 2 | 0
REGURGITATION - MITRAL-INDETERMINATE +3 (Cardiac disorders) | 3 | 0
REGURGITATION - MITRAL-INDETERMINATE +4 (Cardiac disorders) | 3 | 1
REGURGITATION - TRICUSPID-CENTRAL/TRANSVALVULAR +3 (Cardiac disorders) | 1 | 0
REGURGITATION - TRICUSPID-CENTRAL/TRANSVALVULAR +4 (Cardiac disorders) | 4 | 0
REGURGITATION - TRICUSPID-INDETERMINATE +3 (Cardiac disorders) | 2 | 0
REGURGITATION - TRICUSPID-INDETERMINATE +4 (Cardiac disorders) | 2 | 0
STENOSIS - MITRAL - SEVERE (Cardiac disorders) | 1 | 0
THROMBOEMBOLIC EVENT - OTHER - CENTRAL - NO PARESIS (Cardiac disorders) | 1 | 0
THROMBOEMBOLIC EVENT - STROKE (Cardiac disorders) | 56 | 6
THROMBOEMBOLIC EVENT - TRANSIENT ISCHEMIC ATTACK (TIA) (Cardiac disorders) | 27 | 1
VALVE THROMBOSIS - AORTIC (Cardiac disorders) | 1 | 0
HEARING DISORDER (Ear and labyrinth disorders) | 3 | 0
ENDOCRINE COMPLICATIONS (Endocrine disorders) | 4 | 0
PANCREATIC COMPLICATION (Endocrine disorders) | 15 | 0
VISION DISORDER (Eye disorders) | 35 | 0
GASTROINTESTINAL - INFECTION (Gastrointestinal disorders) | 17 | 1
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 108 | 3
ALLERGIC REACTION - MEDICATION RELATED (General disorders) | 2 | 0
ALLERGIC REACTION - OTHER (General disorders) | 1 | 0
ANAPHYLACTIC REACTION (General disorders) | 1 | 0
CANCER - NEWLY DIAGNOSED (General disorders) | 77 | 1
CANCER - PROGRESSION OF UNDERLYING DISEASE (General disorders) | 18 | 1
FEVER - UNKNOWN ORIGIN (General disorders) | 10 | 0
MULTI-SYSTEM ORGAN FAILURE (General disorders) | 8 | 0
NONSPECIFIC, UNKNOWN, OR OTHER BODY SYSTEM - OTHER COMPLICATION (General disorders) | 150 | 7
NSD - PARAVALVULAR LEAK +2 (General disorders) | 2 | 0
NSD - PARAVALVULAR LEAK +3 (General disorders) | 8 | 0
NSD - PARAVALVULAR LEAK +4 (General disorders) | 2 | 1
NSD - PARAVALVULAR LEAK WITH HEMOLYSIS (General disorders) | 2 | 0
NSD - STUDY VALVE STENOSIS - SEVERE (General disorders) | 9 | 0
SPEECH DISORDER (General disorders) | 1 | 0
SVD - STUDY VALVE CALCIFICATION (General disorders) | 5 | 0
BILIARY (GALLBLADDER) (Hepatobiliary disorders) | 29 | 1
HEPATIC COMPLICATION - OTHER (Hepatobiliary disorders) | 4 | 0
LIVER FAILURE - ACUTE (Hepatobiliary disorders) | 1 | 0
INFECTION/INFLAMMATION - OTHER (Infections and infestations) | 49 | 2
STERNAL WOUND/THORACIC INFECTION (Infections and infestations) | 11 | 1
WOUND INFECTION - OTHER (Infections and infestations) | 31 | 0
METABOLIC COMPLICATIONS (Metabolism and nutrition disorders) | 4 | 1
BONE FRACTURE/BREAK (Musculoskeletal and connective tissue disorders) | 57 | 3
MUSCULAR SKELETAL/DERMATOLOGIC - OTHER (Musculoskeletal and connective tissue disorders) | 177 | 4
PSYCHIATRIC - OTHER (Psychiatric disorders) | 20 | 0
PSYCHIATRIC DISORDER (Psychiatric disorders) | 6 | 0
SUICIDE (Psychiatric disorders) | 1 | 0
GENITOURINARY - OTHER (Renal and urinary disorders) | 31 | 1
RENAL - OTHER (Renal and urinary disorders) | 33 | 1
RENAL DYSFUNCTION (Renal and urinary disorders) | 12 | 0
RENAL FAILURE - ACUTE (Renal and urinary disorders) | 41 | 3
RENAL FAILURE - CHRONIC (Renal and urinary disorders) | 3 | 0
URINARY TRACT INFECTION (UTI) (Renal and urinary disorders) | 43 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
HYPOXEMIA (Respiratory, thoracic and mediastinal disorders) | 13 | 0
PLEURAL EFFUSION - BILATERAL (Respiratory, thoracic and mediastinal disorders) | 28 | 0
PLEURAL EFFUSION - LEFT (Respiratory, thoracic and mediastinal disorders) | 21 | 2
PLEURAL EFFUSION - RIGHT (Respiratory, thoracic and mediastinal disorders) | 33 | 4
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 11 | 0
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 6 | 1
PULMONARY EMBOLISM - BILATERAL (Respiratory, thoracic and mediastinal disorders) | 7 | 0
PULMONARY EMBOLISM - LEFT (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM - RIGHT (Respiratory, thoracic and mediastinal disorders) | 6 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY/RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 31 | 2
RESPIRATORY DYSFUNCTION/INSUFFICIENCY (Respiratory, thoracic and mediastinal disorders) | 15 | 2
RESPIRATORY FAILURE - ACUTE RESPIRATORY DISTRESS SYNDROME (ARDS) (Respiratory, thoracic and mediastinal disorders) | 8 | 0
RESPIRATORY FAILURE - ASTHMA (Respiratory, thoracic and mediastinal disorders) | 3 | 0
RESPIRATORY FAILURE - COPD (Respiratory, thoracic and mediastinal disorders) | 16 | 0
RESPIRATORY FAILURE - EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE - HEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 0
RESPIRATORY FAILURE - OTHER (Respiratory, thoracic and mediastinal disorders) | 50 | 4
RESPIRATORY FAILURE - PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 34 | 1
RESPIRATORY FAILURE - PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 5 | 1
RESPIRATORY INFECTION - PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 69 | 4
RESPIRATORY INFECTION - UPPER (URI) (Respiratory, thoracic and mediastinal disorders) | 17 | 0
VASCULAR - ACCESS SITE COMPLICATION (Vascular disorders) | 4 | 0
VASCULAR - DEEP VEIN THROMBOSIS (DVT) (Vascular disorders) | 15 | 1
VASCULAR - OTHER (Vascular disorders) | 44 | 0
PERFORATION - OTHER (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Edwards TRANSFORM INTUITY Aortic Valve Study Cohort (N=885) | Commercially Available Aortic Valve Study Cohort (N=49)
THROMBOCYTOPENIA - NON-HEPARIN INDUCED (Blood and lymphatic system disorders) | 442 | 28
BLOOD/LYMPHATIC - OTHER (Blood and lymphatic system disorders) | 259 | 3
ANEMIA - BLEEDING RELATED - MINOR (Blood and lymphatic system disorders) | 196 | 10
ANEMIA - NON-BLEEDING RELATED (Blood and lymphatic system disorders) | 83 | 9
ARRHYTHMIA - PAROXYSMAL ATRIAL FIBRILLATION (PAF) (Cardiac disorders) | 262 | 15
ARRHYTHMIA - BUNDLE BRANCH BLOCK - LEFT (Cardiac disorders) | 279 | 9
ARRHYTHMIA - AV BLOCK - 1ST DEGREE (Cardiac disorders) | 232 | 11
ARRHYTHMIA - OTHER (Cardiac disorders) | 248 | 12
ARRHYTHMIA - BRADYCARDIA (Cardiac disorders) | 137 | 5
ARRHYTHMIA - BUNDLE BRANCH BLOCK - RIGHT (Cardiac disorders) | 92 | 6
HYPOTENSION (Cardiac disorders) | 161 | 6
CARDIOVASCULAR - OTHER (Cardiac disorders) | 154 | 3
HYPERTENSION - SYSTEMIC (Cardiac disorders) | 80 | 1
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 137 | 5
URINARY TRACT INFECTION (UTI) (Renal and urinary disorders) | 105 | 7
MUSCULAR SKELETAL/DERMATOLOGIC - OTHER (Musculoskeletal and connective tissue disorders) | 234 | 8
NONSPECIFIC, UNKNOWN, OR OTHER BODY SYSTEM - OTHER COMPLICATION (General disorders) | 253 | 8
PSYCHIATRIC - OTHER (Psychiatric disorders) | 77 | 3
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 348 | 14
PLEURAL EFFUSION - BILATERAL (Respiratory, thoracic and mediastinal disorders) | 63 | 1
ENDOCRINE COMPLICATIONS (Endocrine disorders) | 61 | 1
RENAL DYSFUNCTION (Renal and urinary disorders) | 61 | 3
RENAL - OTHER (Renal and urinary disorders) | 59 | 2
RENAL FAILURE - ACUTE (Renal and urinary disorders) | 57 | 1
INFECTION/INFLAMMATION - OTHER (Infections and infestations) | 88 | 4
BONE FRACTURE/BREAK (Musculoskeletal and connective tissue disorders) | 54 | 1
VASCULAR - OTHER (Vascular disorders) | 57 | 2
PULMONARY/RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 108 | 3
RESPIRATORY INFECTION - UPPER (URI) (Respiratory, thoracic and mediastinal disorders) | 60 | 3
THROMBOCYTOPENIA - HEPARIN INDUCED (HIT) (Blood and lymphatic system disorders) | 12 | 3
ARRHYTHMIA - ATRIAL FLUTTER (Cardiac disorders) | 44 | 3
ARRHYTHMIA - PERSISTENT ATRIAL FIBRILLATION (Cardiac disorders) | 38 | 3
ARRHYTHMIA - TACHYCARDIA - NON-VENTRICULAR (Cardiac disorders) | 36 | 4
HEART FAILURE - ACUTE (Cardiac disorders) | 29 | 4
PERICARDITIS (Cardiac disorders) | 13 | 3
GENITOURINARY - OTHER (Renal and urinary disorders) | 35 | 4
VISION DISORDER (Eye disorders) | 47 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can't publish/present on overall study results not yet published but may publish his own data subject to EW review prior to submission/presentation, but data analyses of site-specific results can occur only in intervals as specified in the CTA. Publication/presentation of the PI's site-specific results of devices which haven't been market released and which still may be undergoing development, shall not include claims of device safety/effectiveness and will require the review/approval of EW.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT01700439/Prot_SAP_000.pdf